CLINICAL TRIAL: NCT05813587
Title: A Randomized, Double-blind, Placebo-controlled, Loaded Phase III Clinical Trial on the Efficacy and Safety of Mepozumab for Injection in the Treatment of Post-COVID-19
Brief Title: To Evaluate the Safety and Efficacy of Meplazumab in Treatment of Post-COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Pacific Meinuoke Bio Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPZ-III-02
Record Dates: First submitted 2023-04-10; First posted 2023-04-14 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-02

CONDITIONS: Post-COVID-19
MeSH Terms: interventions — meplazumab; Injections; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meplazumab (Experimental): First dose: 0.2 mg/kg - Day 1; second dose: 0.2 mg/kg - Day 8
  Interventions: Biological: Meplazumab for injection
- Placebo (Placebo Comparator): First dose: control - Day 1; second dose: control - Day 8
  Interventions: Other: Normal saline

INTERVENTIONS:
Biological: Meplazumab for injection — Meplazumab is a humanized anti-CD147 immunoglobulin 2 (IgG2) monoclonal antibody which is expected to block the binding of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spike protein to the human host-cell-expressed CD147, thereby blocking entry of SARS-CoV-2 into human tissue. This expectation is based on in vitro functional studies using Vero E6 cells infected with SARS-CoV-2 that demonstrated effective meplazumab mediated virus gene copy number inhibition upwards of 90% as evaluated by quantitative polymerase chain reaction. Meplazumab may also inhibit COVID-19 associated cytokine storm syndrome based on inhibition of the pro inflammatory factor Cyclophilin A host-cell CD147 interaction.
  Arms: Meplazumab
Other: Normal saline — Normal saline
  Arms: Placebo

SUMMARY:
This trial was a randomized, double-blind, placebo-controlled, loading phase III clinical study.

DETAILED DESCRIPTION:
This test is in the new type of coronavirus infection therapy and 10 (trial version) "and" new coronavirus pneumonia antiviral drug clinical trial technical guidelines (try out) ", on the basis of according to the results of the phase I and phase II clinical study to set up an experimental group and a placebo group, experimental group on the basis of medicines for load test, The control group was loaded with placebo as the base treatment. A planned cohort of 144 patients with Post-COVID-19 (120 +20% dropped out) was randomly assigned in a 1:1 ratio to the experimental group or the placebo group. Mepozumab or placebo was intravenously infused at a dose of 0.2 mg/kg on day 1 (D0). If the clinical symptoms of Post-COVID-19 were not relieved (remission was defined as a decrease in the Post-COVID-19 composite score for at least 2 days), an additional dose of 0.2 mg/kg was administered on day 7 after the first dose, and the actual dose was calculated according to the body weight of the subject. The participants were asked to record the clinical symptoms of Post-COVID-19 daily during the trial. The absent clinical symptoms were evaluated as "zero (none)", and the present clinical symptoms were recorded until they returned to normal (score: zero), which lasted for at least 2 days. On the 28th day (D28±3) after the first dose, the subjects were required to return to the study center again, return their diary cards, and complete each exit examination. If a participant stops the trial early for various reasons, laboratory testing is required to complete the efficacy and safety assessment. During the trial, the subjects were treated according to the type and severity of adverse events according to the clinical diagnosis and treatment standards.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 84 (including 18 and 84), male and female
2. Patients had been infected with 2019-ncov and had at least one symptom of Post-COVID-19 after infection, such as insomnia, memory loss, smell change, taste change, fatigue or fatigue, headache, chest pain, muscle/joint pain, shortness of breath, cough, palpitation, arrhythmia, and aggravation of the primary disease
3. According to the Post-COVID-19 Clinical symptom assessment form , the total symptom assessment score of the subjects was ≥2 before randomization
4. Agree to use highly effective birth control within 3 months of using the experimental drug
5. The subjects were able to communicate well with the investigators, understand and comply with the requirements of the study, and understand and sign the informed consent

Exclusion Criteria:

1. Patients with allergic constitution and known allergic to the test drug and its components

2. Patients who underwent surgery or chemotherapy or radiotherapy within 28 days before screening

3. Patients had a serious systemic disease, condition, or disorder, etc., that was deemed by the investigator to be inappropriate for participation in the study

4. Use of an anti-coronavirus treatment such as Paxlovid (nematavir/ritonavir packaged in combination) within three half-lives before the first dose or during the study period, About 18 h at t1/2), Azvudine tablets (about 9 h at t1/2), and monolavir capsules (about 3.3 h at t1/2) h), ambavirumab/romisivir injection (t1/2 about 45 days /75 days), COVID-19 human immunoglobulin (t1/2 about 3-4 weeks) or recovery plasma (t1/2 about 21 days), deuremidvir hydrobromide tablets (t1/2 about 4.80-6.95 hours), etc

5. At the time of screening, any of the laboratory test indicators meet the following criteria

1. ALT or AST >3ULN
2. Total bilirubin ≥2 ULN
3. White blood cell count > 2 ULN
4. Neutrophil absolute value<0.5×109/L
5. Platelet count < 80×109/L
6. eGFR <60 mL/min/1.73 m2 (calculated by CKD-EPI formula)

Note: For patients with connective tissue diseases such as systemic lupus erythematosus, Sjogren's syndrome, and inflammatory myopathy, including but not limited to the above three diseases, the value of this index was determined by the investigator

6. Weight ≤40 kg

7. Dizzy with needles and blood

8. Had participated in other drug clinical trials within 3 months before screening

9. Pregnant, lactating women or those with a positive pregnancy

10. Other factors that the investigators considered inappropriate for trial entry

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
During the trial (28 days), the duration/degree of relief/recovery of four types of clinical symptoms of Post-COVID-19 | Day28
  The clinical symptoms of Post-COVID-19 mainly involved the nervous system and physical ability (insomnia, memory loss, olfactory changes, taste changes, fatigue or fatigue, headache, chest pain, muscle/joint pain), respiratory system (shortness of breath, cough), cardiovascular system (palpitation, arrhythmia), and aggravation of primary diseases. Clinical symptoms/restore definition: new crown sequela comprehensive score decline, and continue for at least 2 days. Patients with the above symptoms were evaluated according to the actual clinical symptoms, and the clinical symptoms that did not appear were evaluated as "0 (none)"

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of the Air Force Medical University, Xi'an, China